CLINICAL TRIAL: NCT05177861
Title: The Effect of Ulnar Nerve Injury Localization on Sleep Quality in Patients With Ulnar Nerve Entrapment Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator, Yuzuncu Yil University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 100th year University Van
Record Dates: First submitted 2021-12-13; First posted 2022-01-05 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Ulnar Neuropathies
MeSH Terms: conditions — Ulnar Neuropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electromyelography (Other): EMG will be performed only once to determine the ulnar nerve entrapment site in patients.
  Interventions: Diagnostic Test: EMG

INTERVENTIONS:
Diagnostic Test: EMG — Electromyelography

SUMMARY:
Regardless of the cause of ulnar nerve entrapment neuropathy, we are planning to investigate the relationship between sleep quality disorder that may develop due to ulnar neuropathy and the level of entrapment in electromyelography.

ELIGIBILITY:
Inclusion Criteria:

* having ulnar nerve entrapment neuropathy with clinical examination and EMG (electroneuromyography)
* to be between the ages of 18-65
* be give informed consent

Exclusion Criteria:

* malignancy
* surgical history in the ipsilateral upper extremity
* sleep apnea
* narcolepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index | 10 minutes.
  sleep evaluation between 0 and 21 points, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Şah, Principal Investigator — Yüzüncü Yıl Üniversitesi Tıp Fakültesi
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No